CLINICAL TRIAL: NCT03523858
Title: An Open-Label, Single-Arm 4-Year Study to Evaluate Effectiveness and Safety of Ocrelizumab Treatment in Patients With Progressive Multiple Sclerosis
Brief Title: A Study to Evaluate Ocrelizumab Treatment in Participants With Progressive Multiple Sclerosis
Acronym: CONSONANCE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MN39159; 2017-001313-93 (EudraCT Number); 2023-506429-13-00 (EU CTIS Number)
Record Dates: First submitted 2018-04-16; First posted 2018-05-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Progressive Multiple Sclerosis (PMS)
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — ocrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ocrelizumab (Experimental): Ocrelizumab will be administered via intravenous (IV) infusion.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab will be administered via intravenous (IV) infusion at an initial dose of two 300-mg infusions separated by 14 days (on Days 1 and 15), and then 600 mg at every subsequent dose every 24 weeks for the remainder of the study treatment period (approximately 192 weeks)

SUMMARY:
This study is a prospective, multicenter, open-label, single-arm effectiveness and safety study in participants with progressive multiple sclerosis (PMS).

ELIGIBILITY:
Inclusion Criteria:

* Have a definite diagnosis of PMS (as per the revised McDonald 2010 criteria for PPMS or Lublin et al. 2014 criteria for PMS)
* EDSS (Expanded Disability Status Scale) </ =6.5 at screening
* Have a documented evidence of disability progression independent of relapse at any point over the 2 years prior to the screening visit. In case relapse(s) have occurred in the last 2 years, disability progression will have to be considered as independent of relapse activity as per treating physician's judgment
* Fulfill at least one of the 21 criteria assessing the evidence of disability progression independent of relapse activity in the last 2 years using the pre-baseline disability progression rating system checklist
* Have experience of having used a smartphone and connecting a smartphone to Wi-Fi network providers
* For women of childbearing potential: agreement to remain abstinent or use acceptable contraceptive methods during the treatment period and for at least 6 months, or longer if the local label is more stringent after the last dose of study drug

Exclusion Criteria:

* Relapsing-remitting multiple sclerosis (RRMS) at screening
* Inability to complete an MRI
* Gadolinium (Gd) intolerance
* Known presence of other neurological disorders

Exclusions Related to General Health:

* Pregnancy confirmed by positive serum β human chorionic gonadotropin (hCG) measured at screening
* Lactation
* Any concomitant disease that may require chronic treatment of systemic corticosteroids or immunosuppressants during the course of the study
* History or currently active primary or secondary immunodeficiency
* Lack of peripheral venous access
* Significant or uncontrolled somatic disease or any other significant disease that may preclude participant from participating in the study.
* Active infections must be treated and resolved prior to the first infusion of ocrelizumab
* Participants in a severely immunocompromised state until the condition resolves
* Participants with known active malignancies or being actively monitored for recurrence of malignancy
* Participants who have or have had confirmed progressive multifocal leukoencephalopathy (PML)

Exclusions Related to Laboratory Findings:

* Positive screening tests for hepatitis B
* CD4 count <250/μL
* ANC <1.0 × 103/μL
* AST/SGOT or ALT/SGPT ≥3.0 × ULN in combination with either an elevated total bilirubin (>2 X ULN) or clinical jaundice

Exclusions Related to Medications:

* Hypersensitivity to ocrelizumab or to any of its excipients
* Previous treatment with ocrelizumab
* Previous treatment with B-cell targeted therapies (i.e., atacicept, tabalumab, belimumab, ofatumumab, or obinutuzumab). Note: previous treatment with rituximab is allowed as long as the last dose was administered more than 6 months before the ocrelizumab infusion AND if discontinuation was due to adverse events or immunogenicity AND if Bcell levels are above the lower limit of normal (LLN) prior to screening.
* Any previous treatment with alemtuzumab (Campath/Mabcampath/Lemtrada), total body irradiation, or bone marrow transplantation
* Previous treatment with natalizumab where PML has not been excluded according to specific algorithm
* Contraindications to or intolerance of oral or intravenous (IV) corticosteroids, including methylprednisolone administered IV, according to the country label
* Systemic corticosteroid therapy within 4 weeks prior to screening
* All vaccines should be given at least 6 weeks before the first infusion of ocrelizumab, unless the local regulations allow for a shorter interval. Live/live attenuated vaccines should be avoided during treatment and safety follow-up period until B cells are peripherally repleted
* Previous treatment with daclizumab, ozanimod or figolimod in the last 8 weeks
* Previous treatment with siponimod in the last 2 weeks
* Treatment with fampridine/dalfampridine (Fampyra)/Ampyra) or other symptomatic MS treatment unless on stable dose for ≥30 days prior to screening
* Previous treatment with natalizumab in the last 12 weeks.
* Previous treatment with teriflunomide in the last 12 weeks. This washout period can be shortened if an accelerated elimination procedure is implemented before screening visit. One of the following elimination procedures can be used:
* Cholestyramine 8 g administered 3 times daily for a period of at least 7 days (cholestyramine 4 g three times a day can be used, if cholestyramine 8 g three times a day is not well tolerated)
* Alternatively, 50 g of activated powdered charcoal is administered every 12 hours for a period of at least 7 days.
* Previous treatment with azathioprine, cyclophosphamide, mycophenolate mofetil or methotrexate in the last 12 weeks
* Treatment with any investigational agent within 24 weeks of screening (Visit 1) or five half-lives of the investigational drug (whichever is longer) or treatment with any experimental procedures for MS
* Previous treatment with mitoxantrone, cyclosporine or cladribine in the last 96 weeks
* Participants previously treated with teriflunomide within the last two years, unless measured plasma concentrations are less than 0.02 mg/l. If above or not known, an accelerated elimination procedure should be implemented before screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2026-11-12 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with No Evidence of Progression (NEP) | From Baseline to Week 96, Week 96 to Week 192 and Baseline to Week 192
  NEP is defined as no progression sustained for at least 24 weeks on all of the following three components (confirmed disability progression [CDP]; ≥20% increase in timed 25-foot walk test [T25FWT]; ≥20% increase in nine-hole peg test [9HPT])
Proportion of Participants with no evidence of progression and no active disease (NEPAD) | From Baseline to Week 96, Week 96 to Week 192 and Baseline to Week 192
  NEPAD is defined as no progression sustained for at least 24 weeks on all of the three components of NEP (CDP, T25FWT, 9HPT), no protocol-defined relapse, no enlarging or new T2 lesion, and no T1 gadolinium (Gd+)-enhancing lesion

SECONDARY OUTCOMES:
Change from Baseline in Cognitive Function, as Measured by the Symbol Digit Modalities Test (SDMT) | Baseline to end of study (Week 192)
Change from Baseline in Cognitive Function, as Measured by Brief Visuospatial Memory Test - Revised (BVMT-R) | Baseline to end of study (Week 192)
Mean Change from Baseline in the Expanded Disability Status Scale (EDSS) score over the course of the study | Baseline to end of study (Week 192)
Time to Onset of First Confirmed Disability Progression (CDP) Sustained for at least 24 and 48 Weeks | Baseline to onset of first CDP (as measured by EDSS) sustained for at least 24 and 48 weeks
Time to Onset of First >=20% Increase in Timed 25-foot Walk Test (T25FWT) Sustained for at least 24 Weeks | Baseline to onset of first >=20% increase in T25FWT sustained for at least 24 weeks
Time to Onset of First >=20% Increase in 9 Hole Peg Test (9HPT) Sustained For At Least 24 Weeks | Baseline to onset of first >=20% increase in 9HPT sustained for at least 24 weeks
Proportion of Participants with NEP | Week 24 to Week 96, Week 24 to Week 192, and Week 48 to Week 192
Proportion of Participants with NEPAD | Week 24 to Week 96, Week 24 to Week 192, Week 48 to Week 192
Change from Baseline in Patient-Reported Outcomes (PROs) | Baseline to end of study (Week 192)
  PROs collected in this study will be the Multiple Sclerosis Impact Scale (MSIS-29), the Multiple Sclerosis Walking scale (MSWS-12), the ABILHAND-56 Questionnaire, Fatigue Scale for Motor and Cognitive function (FSMC), SymptoMScreen, 88-item Multiple Sclerosis Spasticity Scale (MSSS-88), Numerical Pain Rating Scale (NPRS), and the Patient Global Impression of Severity (PGIS) for upper limb, lower limb and cognitive function
Change from Baseline in the number of falls and near-falls | Baseline to end of study (Week 192)
Change in Whole Brain Volume (Whole, Cerebral White Matter, Cortical Grey Matter, Deep grey matter) | Baseline to end of study (Week 192)
Change in thalamic volumes | Baseline to end of study (Week 192)
Change in whole and regional cerebellar volume (cervical cord grey and white matter area) | Baseline to end of study (Week 192)
Change in cervical cord cross-sectional area (total, white matter and grey matter) | Baseline to end of study (Week 192)
Change in number of new/enlarging T2 lesions and total T2 Lesion Volume | Baseline to end of study (Week 192)
Change in number of T1 Gadolinium (Gd)+ Lesions and total volume | 'Baseline to end of study (Week 192)
Change in number of T1 lesions | Baseline to end of study (Week 192)
Number in total volume of T1 lesions | Baseline to end of study (Week 192)
Change in Slowly Evolving Lesions (SEL) | Baseline to end of study (Week 192)
Change in normalised T1 intensity/T1 Gd+ enhancement in New Focal T2 Lesions, SELs, Persistent Areas of Non-SEL T2 Lesions, and Normal-Appearing Brain Tissue | Baseline to end of study (Week 192)
Change in Gd-enhancing late-Fluid-Attenuated Inversion-Recovery (FLAIR) Meningeal Lesions | Baseline to end of study (Week 192)
Change in the number/ spatial distribution of lesions in the cervical spinal cord | Baseline to end of study (Week 192)
Spectroscopic MR: Measure of the Relative Signal Amplitude of N-Acetyl Aspartate (NAA), and Choline to Creatine | Baseline to end of study (Week 192)
  Only in centers with 1.5-Tesla MRI capable to perform it
Measure of phase rim lesions using a Susceptibility-Weighted Imaging [SWI]/T2 sequence | Baseline to end of study (Week 192)
  Only in centers with 3-Tesla MRI capable to perform it, where this sequence would replace the spectroscopic MR in the acquisition flow
Percentage of Participants with Adverse Events (AEs) | Baseline to end of study (Week 192)
Rates of study treatment discontinuation due to adverse events | Baseline to Week 192

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (124):
- United States (18):
  - MS Center of California, Laguna Hills, California
  - SC3 Research Group, Inc, Pasadena, California
  - University of California San Francisco, San Francisco, California
  - Yale University, North Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dragonfly Research, LLC, Wellesley, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - The MS Center of Northeastern New York, Latham, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Mellen Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Neurology Clinic PC, Cordova, Tennessee
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Lone Star Neurology of San Antonio, San Antonio, Texas
  - Swedish Multiple Sclerosis Center, Seattle, Washington
- Bosnia and Herzegovina (4):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - University Hospital Mostar, Mostar
  - Clinical Center University of Sarajevo, Sarajevo
  - University Clinical Center Tuzla, Tuzla
- Brazil (4):
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas Faculdades Médicas de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Hospital das Clinicas - FMUSP_X, São Paulo, São Paulo
- Canada (7):
  - Fraser Health Authority - Fraser Health Multiple Sclerosis, Burnaby, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia
  - London Health Sciences Centre Uni Campus, London, Ontario
  - St. Michael'S Hospital, Toronto, Ontario
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Hospital Notre-Dame du Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
- Colombia (2):
  - Organizacion Sanitas Internacional, Bogotá
  - Fundacion Clinica Valle del Lili, Cali
- Hospital Clínica Biblica, San José, Costa Rica
- Czechia (4):
  - Nemocnice Jihlava, Jihlava
  - Fakultní Nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, Glostrup Municipality
  - Hjerne- og nervesygdomme, Ambulatorium, Skleroseklinikken, Sønderborg
- Egypt (2):
  - Clinical Research Center-Alex university, Alexandria
  - Neurology Department, Ain Shams University Hospitals, Cairo
- France (15):
  - CHIC Cote Basque Bayonne, Bayonne
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital neurologique Pierre Wertheimer - CHU Lyon, Bron
  - CHU De Caen, Caen
  - Hopital Gabriel Montpied CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hopital B Roger Salengro, Lille
  - CHU de la Timone - Hopital d Adultes, Marseille
  - Hopital Gui de Chauliac, Montpellier
  - CHRU Nancy, Nancy
  - Hopital Nord Laennec, Nantes
  - Hôpital Pasteur, Nice
  - GroupeHospitalo-Universitaire Caremeau, Nîmes
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - CHU Amiens Hopital Sud, Salouël
  - Hopitaux Universitaires de Strasbourg, Strasbourg
- Germany (6):
  - Universitätsklinikum "Carl Gustav Carus", Zentrum für Klinische Neurowissenschaften, Dresden
  - Universitätsmedizin Greifswald, Greifswald
  - NeuroConcept AG C/O mind mvz GmbH, Stuttgart
  - NeuroPoint Gesellschaft fur vorbeugende Gesundheitspflege mbH, Ulm
  - Studienzentrum Nordwest Dr med Joachim Springub Herr Wolfgang Schwarz, Westerstede
  - Deutsche Klinik für Diagnostik, Wiesbaden
- Nucare, Guatemala City, Guatemala
- Hungary (4):
  - Semmelweis Egyetem AOK, Budapest
  - VALEOMED Diagnosztikai Központ, Esztergom
  - Jósa András Oktatókórház, Nyíregyháza
  - Pécsi Tudományegyetem, Klinikai Központ Neurológiai Klinika, Pécs
- Ireland (3):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St Vincents University Hospital, Dublin
- Italy (20):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di, Bari, Apulia
  - A. O. U. Federico II, Napoli, Campania
  - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Università degli studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Ospedale Cattinara, Trieste, Friuli Venezia Giulia
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - Policlinico Universitario A. Gemelli, Rome, Lazio
  - A.O. Sant'Andrea, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Irccs A.O.U.San Martino Ist, Genoa, Liguria
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Fond. Istituto Neurologico C.Besta, Milan, Lombardy
  - IRCCS Istituto Neurologico C. Mondino?Dip. Neurologia Neuroriabilitazione S.S. Sclerosi Multipla, Pavia, Lombardy
  - IRCCS Istituto Neurologico Neuromed, Pozzilli, Molise
  - Azienda Sanitaria Ospedaliera S. Luigi Gonzaga, Orbassano, Piedmont
  - AOU Città della Salute e della Scienza, Turin, Piedmont
  - Ospedale Binaghi, Cagliari, Sardinia
  - AOU Policlinico V. Emanuele - P.O G. Rodolico, Catania, Sicily
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Policlinico G.B. Rossi, Verona, Veneto
- Lebanon (2):
  - American University of Beirut - Medical Center, Beirut
  - Lebanese American University Medical Center- Rizk Hospial, Beirut
- Mexico (4):
  - Grupo Medico de Investigacion Clinica Multidisciplinaria, Mexico City, Mexico CITY (federal District)
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - Hospital General de Mexico, Mexico, Tlaxcala
  - Unidad de investigacion en salud (UIS), Mexico City
- Morocco (3):
  - Centre Hospitalier Universitaire Hassan II, Fes
  - Hopital Cheikh Zaid, Rabat
  - Hopital Militaire d'Instruction Mohamed V, Rabat
- Netherlands (4):
  - Amphia Ziekenhuis, Breda
  - Catharina ziekenhuis, Eindhoven
  - Maasstadziekenhuis, NL -rotterdam
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
- Consultorios Médicos PaItilla, Panama City, Panama
- Poland (7):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - SP Swiecickiego UM Marcinkowskiego, Późna
  - Centrum Medyczne "MEDYK", Rzeszów
  - Wojskowy Instytut Medyczny - Pa?Stwowy Instytut Badawczy, Warsaw
  - SPSK nr 1, Zabrze
- Russia (4):
  - Jusupovskaya Hospital, Moscow, Moscow Oblast
  - Vladimirskiy Regional Scientific Research Inst., Moscow, Moscow Oblast
  - City Clinical Hospital #24, Moskva, Moscow Oblast
  - National Center of Social Significant Disease, Saint Petersburg, Sankt-Peterburg
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital Universitario la Fe, Valencia
- United Arab Emirates (2):
  - Cleveland Clinic Abu Dhabi, Abu Dhabi
  - Rashid hospital, Dubai

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Kappos L, Yiu S, Dahlke F, Coetzee T, Cutter GR, Yuen S, Bonati U, Lublin FD. Composite Confirmed Disability Worsening/Progression Is a Useful Clinical Endpoint for Multiple Sclerosis Clinical Trials. Neurology. 2025 May 27;104(10):e213558. doi: 10.1212/WNL.0000000000213558. Epub 2025 Apr 21. PMID 40258203